CLINICAL TRIAL: NCT00368940
Title: A Treatment for Depressed, Cognitively Impaired Elders
Brief Title: Problem Adaptation Therapy (PATH) vs. Supportive Therapy in Treating Depressed, Cognitively Impaired Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23MH074659 (NIH); K23MH074659 (NIH); 0301005971; DATR AK-TNGP2
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-04

CONDITIONS: Depression
Keywords: Memory Deficits; Geriatric Depression; Cognitive Impairment; Executive Dysfunction; Disability; Problem Solving Therapy
MeSH Terms: conditions — Depression; Memory Disorders; Cognitive Dysfunction | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PATH (Experimental): Participants will receive PATH for 12 weeks
  Interventions: Behavioral: PATH
- ST-CI (Active Comparator): Participants will receive ST-CI for 12 weeks
  Interventions: Behavioral: ST-CI

INTERVENTIONS:
Behavioral: PATH — PATH utilizes a problem solving approach based on Problem Solving Therapy (PST) and identifies problems that interfere with everyday functions and that contribute to depression and disability. The treatment then provides compensatory strategies and environmental adaptations that are designed to bypass the person's cognitive limitations and to improve adaptive functioning in the home environment. PATH also incorporates caregiver involvement to help patient reduce depression and improve functioning.
  Arms: PATH
Behavioral: ST-CI — Supportive therapy focuses on the use of nonspecific or common factors of therapy, including facilitation of affect, helping the person feel understood, empathy, the treatment ritual, success experiences, and therapeutic optimism. In working with the participant, the therapist creates a supportive relationship and encourages the participant to consider his/her strengths and abilities rather than focusing on negative aspects of his/her character.
  Other Names: Supportive Therapy for Cognitively Impaired Older Adults
  Arms: ST-CI

SUMMARY:
This study will evaluate the efficacy of Problem Adaptation Therapy (PATH) vs. Supportive Therapy for Cognitively Impaired (ST-CI) older adults in reducing depression and disability in treating depressed, cognitively impaired older adults.

DETAILED DESCRIPTION:
Depression, cognitive impairment, and disability often coexist in older adults and can lead to patient suffering and family disruption. Moreover, many depressed, cognitively impaired older adults have slow, poor, or unstable response to antidepressant drugs. Despite the need for treatments other than medication, most psychotherapy research focuses on either cognitively intact patients with limited disability or on dementia patients with pronounced disability. Thus, the available treatments do not fully address the needs of the large number of depressed elders with intermediate cognitive impairment and disability. Previous studies with cognitively impaired psychiatric populations have taught participants compensatory strategies to overcome their behavioral and cognitive limitations. This study will evaluate the efficacy of Problem Adaptation Therapy (PATH) a type of psychotherapy using a problem solving therapy (PST) approach, specially tailored compensatory strategies and environmental adaptations and caregiver involvement in treating depressed, cognitively impaired older adults.

All participants in this single-blind study will undergo initial evaluations, including a 2-hour interview to assess depression, memory, and physical functioning; questions about medical history; and a neuropsychological exam. Participants will then be randomly assigned to one of two treatment groups: PATH or ST-CI. Participants assigned to PATH will receive 12 weekly sessions conducted at the home of the participants. During these sessions, a therapist will identify the participant's difficulties in life related to depression and physical functioning and will provide strategies to overcome these difficulties. The goal of treatment is to improve adaptive functioning in the home environment, which in turn may reduce depression and disability. The first session will last between 1 and 2 hours, and the remaining 11 sessions will last 1 hour. Participants assigned to ST-CI will also receive 12 weekly treatment sessions with a therapist conducted at the home of the participants. During supportive therapy sessions, the therapist will help participants to express feelings and to focus on their strengths and abilities when working through difficulties and transitions. For all participants, initial assessments will be repeated at Weeks 4, 8, 12, and 24.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual for Mental Disorders(DSM)IV criteria for unipolar major depression
* Severity of depression greater than or equal to 17 on MADRS
* Disability as determined by at least 1 impairment in instrumental activities of daily living
* Evidence of executive dysfunction or impairment in at least one of the following cognitive domains of Dementia Rating Scale (DRS): attention, construction, conceptualization, and memory ([scaled score less than 7] adjusted for age and race based on Mayo's older participants normative data)
* Family member or caregiver able and willing to participate in treatment
* Not currently taking antidepressants, cholinesterase inhibitors, or memantine or on a stable dosage for 8 weeks prior to study entry with no medical recommendation for change of these agents in the near future

Exclusion Criteria:

* High suicide risk
* Axis I psychiatric disorder or substance abuse other than unipolar major depression or nonpsychotic depression
* Axis II diagnosis of antisocial personality
* Moderate to severe dementia: DRS total score corresponding to moderate or more severe impairment (scaled score less than or equal to 5)
* Acute or severe medical illness (e.g., delirium; metastatic cancer; decompensated cardiac; liver or kidney failure; major surgery; stroke; myocardial infarction during the 3 months prior to entry)
* Currently taking drugs known to cause depression (e.g., reserpine, alpha-methyl-dopa, steroids)
* Currently receiving psychotherapy
* Aphasia
* Sensory problems
* Inability to speak English

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 74 (Actual)
Dates: Start 2006-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris N. Kiosses, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Cornell Institute of Geriatric Psychiatry, White Plains, New York, United States

REFERENCES:
- [Derived] Kanellopoulos D, Rosenberg P, Ravdin LD, Maldonado D, Jamil N, Quinn C, Kiosses DN. Depression, cognitive, and functional outcomes of Problem Adaptation Therapy (PATH) in older adults with major depression and mild cognitive deficits. Int Psychogeriatr. 2020 Apr;32(4):485-493. doi: 10.1017/S1041610219001716. Epub 2020 Jan 8. PMID 31910916
- [Derived] Arslanoglou E, Banerjee S, Pantelides J, Evans L, Kiosses DN. Negative Emotions and the Course of Depression During Psychotherapy in Suicidal Older Adults With Depression and Cognitive Impairment. Am J Geriatr Psychiatry. 2019 Dec;27(12):1287-1295. doi: 10.1016/j.jagp.2019.08.018. Epub 2019 Aug 26. PMID 31582195
- [Derived] Kiosses DN, Gross JJ, Banerjee S, Duberstein PR, Putrino D, Alexopoulos GS. Negative Emotions and Suicidal Ideation during Psychosocial Treatments in Older Adults with Major Depression and Cognitive Impairment. Am J Geriatr Psychiatry. 2017 Jun;25(6):620-629. doi: 10.1016/j.jagp.2017.01.011. Epub 2017 Jan 19. PMID 28223082
- [Derived] Kiosses DN, Ravdin LD, Gross JJ, Raue P, Kotbi N, Alexopoulos GS. Problem adaptation therapy for older adults with major depression and cognitive impairment: a randomized clinical trial. JAMA Psychiatry. 2015 Jan;72(1):22-30. doi: 10.1001/jamapsychiatry.2014.1305. PMID 25372657

RESULTS

PARTICIPANT FLOW:
Groups:
- PATH: Participants will receive PATH for 12 weeks
  PATH: PATH aims to improve emotion regulation and reduce the negative impact of behavioral and functional limitations. The strategies of PATH are consistent with the process model of emotion regulation. PATH utilizes a problem solving approach based on Problem Solving Therapy (PST) and identifies problems that interfere with everyday functions and that contribute to depression and disability. The treatment then provides compensatory strategies and environmental adaptations that are designed to bypass the person's cognitive limitations and to improve adaptive functioning in the home environment. PATH also incorporates caregiver involvement to help patient reduce depression and improve functioning.
Period: Intention-to-Treat
Arm/Group | PATH | ST-CI
Started | 37 | 37
Completed | 37 | 37
Not Completed | 0 | 0
Period: Completed 12-wk Treatment
Arm/Group | PATH | ST-CI
Started | 37 | 37
Completed | 31 | 32
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PATH | ST-CI | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 37 | 37 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 34 | 37 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 30 | 31 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 37 | 74

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Scale (MADRS)
Description: Montgomery Asberg Depression Scale (MADRS) is a depression rating scale. Range of scores (1-35). Higher scores represent worse outcome (depression).
Time Frame: 12 week outcome
Measure: Least Squares Mean (Standard Error); unit: Units on MADRS scale
Arm/Group | PATH | ST-CI
Number analyzed (Participants) | 37 | 37
Units on MADRS scale | 10.46 (1.07) | 15.53 (1.07)
Statistical Analysis 1: Comparison: PATH vs ST-CI; Test type: Superiority; p = 0.005, Mixed Models Analysis; Cohen D at week 12 = 0.60, 95% CI 2-sided [0.13 to 1.06]

2. Primary Outcome: WHO Disability Assessment Schedule (WHODAS)-II
Description: WHO Disability Assessment Schedule (WHODAS)-II is a disability scale. Range of scores: 12-43. Higher scores represent worse outcome (disability).
Time Frame: 12-week outcome
Measure: Least Squares Mean (Standard Error); unit: WHODAS-II units
Arm/Group | PATH | ST-CI
Number analyzed (Participants) | 37 | 37
WHODAS-II units | 27.37 (1.16) | 32.14 (1.15)
Statistical Analysis 1: Comparison: PATH vs ST-CI; Test type: Superiority; p = 0.001, Mixed Models Analysis; Cohen D at week 12 = 0.67, 95% CI 2-sided [0.20 to 1.14]

3. Secondary Outcome: Hamilton Depression Rating Scale
Description: Hamilton Depression Rating Scale is a scale measuring depression severity. Range of scores: 1-33. Higher scores reflect worse outcome (depression).
Time Frame: Outcome at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PATH | ST-CI
Number analyzed (Participants) | 30 | 30
units on a scale | 11.16 (6.9) | 15.03 (7.30)
Statistical Analysis 1: Comparison: PATH vs ST-CI; Test type: Superiority; p = 0.0268, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Sheehan Disability Scale.
Description: Sheehan Disability Scale is a measure of disability. Range of scores: 0-20. Higher scores reflect worse outcome (disability).
Time Frame: Outcome at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PATH | ST-CI
Number analyzed (Participants) | 30 | 31
units on a scale | 5.40 (4.91) | 12.16 (3.87)
Statistical Analysis 1: Comparison: PATH vs ST-CI; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From enty to 24 weeks
Arm/Group | PATH | ST-CI
All-Cause Mortality (participants affected / at risk) | 1/37 | 1/37
Serious Adverse Events (participants affected / at risk) | 8/37 | 10/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PATH (N=37) | ST-CI (N=37)
Hospitalization due to a fall (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Tumor removal (Surgical and medical procedures) | 1 (1) | 1 (1)
Hospitalization for COPD or fluid in lungs (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hospitalization due to possible stroke (Vascular disorders) | 1 (1) | 1 (1)
Hospitalization due to stomach virus or ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hospitalization following an exacerbation of scleroderma (Immune system disorders) | 0 (0) | 1 (1)
Cataract Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No